CLINICAL TRIAL: NCT01142076
Title: Xinju Xiaogao Prescription and 10% of it in the Treatment of Adiposity (Stagnation of QI Causing Phlegm Retention)Clinical Study
Brief Title: Xinju Xiaogao Prescription Study on Overweight
Acronym: XJXG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: China-Japan Friendship Hospital (Other); The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Principal Investigator, Fengmei Lian, chief, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19850701
Record Dates: First submitted 2010-05-24; First posted 2010-06-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Overweight
Keywords: adiposity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Dose treatment group, 10%
  Interventions: Drug: placebo
- Xinju Xiaogao Prescription (Active Comparator): treatment group
  Interventions: Drug: Xinju Xiaogao Prescription

INTERVENTIONS:
Drug: Xinju Xiaogao Prescription — treatment group
  Other Names: Xinju Xiaogao decoction
  Arms: Xinju Xiaogao Prescription
Drug: placebo — Therapeutic dose of 10%
  Arms: placebo

SUMMARY:
Xinju Xiaogao prescription and 10% of it in the treatment of adiposity (stagnation of QI causing phlegm retention)clinical study

DETAILED DESCRIPTION:
Charged by the three research centers in line with traditional Chinese medicine stagnation of QI causing phlegm retention 120 cases have diabetes were randomly divided into Chinese herbal compound Xinju Xiaogao prescription group and 10% of the prescription group.The treatment groups were compared 24-week step-down and regulation of body weight,waistline, blood lipids, blood sugar effect.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years old
* BMI≥28kg/m2，but<40kg/m2
* Waistline≥85cm（male）,≥80cm（female）
* Pathoglycemia must fulfill one of those four condition:
* IGT,7.8≤2hPG≤11.0mmol/,
* diabetics take medicine used to treat type 2 diabetes more than 3 month,and 5.6≤FBG≤12.2,and weight change under 4kg.
* stagnation of QI causing phlegm retention
* To sign informed consent.

Exclusion Criteria:

* After 3-6 months simply controlling their diet and more exercise treatment, body weight weight loss ≥ 5%.
* TG>4.5mmol/L.
* Suffering from congenital heart disease, rheumatic heart disease, kidney disease, serious active liver disease, peptic ulcer disease or malabsorption syndrome.
* There is a history of pancreatitis or endocrine diseases other than diabetes, diabetes treated with insulin.
* Not suffered myocardial infarction in Past 3 months or unstable angina were confirmed.
* Had been diagnosed as "post-surgical adhesions" .
* There is a history of appetite or abuse of laxatives
* Diastolic blood pressure,uncontrolled or controlled, three times greater than 105mmHg .
* Pregnancy, prepare to pregnant or lactating women prepare.
* Allergies to Chinese medicine , allergic.
* Recurrent gallstone or a history of kidney stones.
* Mentally ill.
* Cancer patients.
* A history of gastrointestinal surgery to lose weight.
* Receiving other clinical studies nearly 3 months.
* Alcohol and / or psychoactive substances, drug abusers and addicts.
* Taking other weight-reducing aid Close within one month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
waistline | up to 24 weeks

SECONDARY OUTCOMES:
Body Mass Index (BMI) | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fenglian Li, PHD, Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences